CLINICAL TRIAL: NCT06497478
Title: Evolutionary Aspects of Polydistrict Atherosclerosis (EAP). Analysis and Correlation of Functional, Biomolecular and Genetic Factors.
Brief Title: Evolutionary Aspects of Polydistrict Atherosclerosis
Acronym: EAP
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6415
Record Dates: First submitted 2024-07-05; First posted 2024-07-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2014-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonographic examination — Ultrasonographic examination will be performed using a high-resolution (Epiq Elite Philips Medical Systems, Monza, Italia) and a linear 12-9 MHz transducer.
  The patients will be placed in a supine position. Starting with the probe at the base of the neck, the common carotid artery will be explored on the transverse plane and then on the sagittal one, continuing in a cranial sense up to the carotid bifurcation. The medium-intimal thickness will be measured, defined as distance from the first hyperechoic line to the second hyperechoic line.
  The femoropopliteal and run-off segments will be continuously scanned from the subinguinal region to the paramalleolar region with axial and sagittal scans. All segments will be examined for the presence of vessel wall calcifications and/or atherosclerotic plaques. In addition, flow velocity measurements will be obtained using spectral Doppler imaging and color Doppler imaging.

SUMMARY:
Atherosclerosis is a systemic, multifocal disease that represents the leading cause of death in Western countries. The risk factors contributing to its distribution, extent and progression in different organs (i.e., the heart, brain or limbs) and different segments (large and small vessels) are not identical. The present study analyses data the evolutionary aspects of polydistrict atherosclerosis by analysing the possible role of morphological factors, biomolecular and genetic in the progression of atherosclerotic lesions and the development of major and/or minor acute cardiovascular events.

For this purpose, will be recalled to follow-up all 320 patients already enrolled in the previous protocol of Research in the period between 1 March 2014 and 28 February 2015 at the Department of Internal Medicine, Catholic University of Rome.

The subjects will undergo a new clinical evaluation, with particular interest to the onset of major cardiovascular events (myocardial infarction, stroke, death for all causes) and major adverse events to the lower limbs (critical ischemia of the lower limbs requiring revascularization or amputation) in the follow-up period, and a ultrasonographic examination of carotid arteries and arteries of lower limb districts at the Service of Angiology, Catholic University of Rome.

The study employed a new semiquantitative ultrasonographic score (ultrasonographic lower limb atherosclerosis (ULLA) score), that enables a complete evaluation of the entire lower limb atherosclerotic burden and has already been shown to be associated with major cardiovascular risk factors.

Therefore, the aims of this study are:

* to assess the association between functional, morphological, biomolecular and genetic factors of atherosclerotic disease and the risk of major cardiovascular events (MACE) and major adverse events to the lower limbs (MALE);
* to analyse the morphological progression of atherosclerotic disease in its different localizations and the possible determining factors in such progression with a 10-year follow-up ultrasound study.

ELIGIBILITY:
Inclusion Criteria:

* Follow-up of n.320 subjects previously enrolled in the period between 1 March 2014 and 28 February 2015 in the previous Research Protocol at the Department of Internal Medicine, Catholic University of Rome.

Exclusion Criteria:

* Acute diseases;
* Age < 18 years;
* Inclusion in another clinical trial;
* Impossibility of follow-up (homeless, residence abroad)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes males and females, older than 18 years, who go to the the Department of Internal Medicine, Catholic University of Rome for a follow-up visit involving a medical history assessment, an objective examination and the performance of ultrasound examinations. The study previews the recruitment of subjects already gone to the aforementioned department in the period between 1 July 2014 and 30 June 2015. Patients should have symptoms related to peripheral arterial disease of the lower limbs and/or known cardiovascular risk factors, also in the absence of symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Assessment evolutionary aspects of atherosclerosis | 6 months
  The association between functional, morphological, biomolecular and genetic factors of atherosclerotic disease and the risk of major cardiovascular events (MACE) and major adverse events to the lower limbs (MALE)

SECONDARY OUTCOMES:
Morphological progression of atherosclerosis and factors involved | 6 months
  The morphological progression of atherosclerotic disease in its different localizations and the possible determining factors related to such progression assesed by a 10-year follow-up ultrasound study

CONTACTS AND LOCATIONS:
Overall Officials: luca Santoro, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Medicina Interna, Roma, Italy